CLINICAL TRIAL: NCT01207414
Title: A 12-week, Randomized, Multi-center, Open-Label, Iloperidone, (12-24 mg/Day), Flexible Dose Study Assessing Efficacy, Safety and Tolerability of Two Switch Approaches in Schizophrenia Patients Currently Receiving Risperidone, Olanzapine or Aripiprazole
Brief Title: Switching to Iloperidone From Other Antipsychotics in Schizophrenia
Acronym: i-FANS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CILO522DUS01
Record Dates: First submitted 2010-09-19; First posted 2010-09-22 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; iloperidone; switch; gradual switch; immediate switch
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

ARMS (2):
- iloperidone gradual switch (Experimental): Participants taking risperidone, olanzapine or aripiprazole gradually decreased the dose they were taking: 50% of original dose on Day 1, 25% of original dose after the first week and the total discontinuation of the drug after the second week.
  On Day 1 participants began taking iloperidone orally twice a day (bid) in the morning and in the evening beginning at a dose of 1 mg and increasing to 2 mg, 4 mg, 6 mg, 8 mg, 10 mg, and 12 mg bid on consecutive days over a 7-day period to achieve a total dose of 12-24 mg/day for 12 weeks.
  Interventions: Drug: iloperidone
- iloperidone immediate switch (Experimental): Participants taking risperidone, olanzapine or aripiprazole discontinued the drug immediately.
  On Day 1 participants began taking iloperidone orally twice a day (bid) in the morning and in the evening beginning at a dose of 1 mg and increasing to 2 mg, 4 mg, 6 mg, 8 mg, 10 mg, and 12 mg bid on consecutive days over a 7-day period to achieve a total dose of 12-24 mg/day for 12 weeks.
  Interventions: Drug: iloperidone

INTERVENTIONS:
Drug: iloperidone — Iloperidone tablets supplied at doses of 1 mg, 2 mg, 4 mg, 6 mg, 8 mg, 10 mg and 12 mg to achieve a target dose of 12-24 mg/day for 12 weeks.
  Other Names: Fanapt™

SUMMARY:
Evaluate the clinical outcome of two switching strategies to iloperidone treatment in adult subjects with schizophrenia who require a change in their current antipsychotic treatment of risperidone, olanzapine, or aripiprazole due to suboptimal efficacy and/or safety/tolerability reasons.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 64 years of age, inclusive
* DSM-IV diagnosis of schizophrenia
* Patients currently on an optimal in-label dose of one of the following permitted antipsychotic treatments for at least 30 days: risperidone, olanzapine, or aripiprazole
* Efficacy Clinical Global Impression of Severity (E-CGI-S) of 4 or 5 or
* Not tolerating one of the permitted treatments and exhibits one of the allowable side-effects

Exclusion Criteria:

* Any other current Axis I disorder other than schizophrenia which is the focus of treatment;
* Acutely psychotic or patient's symptom severity requires hospitalization
* Patient with significant cardiovascular illness (myocardial infarction, cardiac arrhythmia)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 501 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla Hochfeld, MD, MD, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (59):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - Comprehensive Neuroscience, Cerritos, California
  - ATP Clinical Research Center, Inc., Costa Mesa, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - Pacific Health Systems, National City, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Inc., Oceanside, California
  - University of California, Irvine, Orange, California
  - CNRI San Diego, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Viking Clinical Research, Temecula, California
  - Collaborative Neuroscience, Torrance, California
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Comprenhensive Neuroscience, Washington D.C., District of Columbia
  - Amit K. Vijapura MD & Associates, Jacksonville, Florida
  - Scientific Clinical Research, North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive Neuroscience, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Carman Research, Smyrna, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Alexian Brothers Center for Mental Health, Arlington Heights, Illinois
  - Rush University Medical Center, Treatment Research Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - AMR - Baber Research, Inc., Naperville, Illinois
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Neurobehavioral Medicine Group, Clinical Trials Division, Bloomfield Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRI World Wide Clinical Research Company, Willingboro, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Neurobehavioral Research, Cedarhurst, New York
  - Comprehensive Neuroscience, Fresh Meadows, New York
  - Division of Psychiatry Research - Zucker Hills Hospital, Glen Oaks, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Behavioral Medical Research, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - North Coast Clinical Trials, Beachwood, Ohio
  - Neurobehavioral Clinical Research, Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - CRI Worldwide, LLC - Kirkbride Division, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Charleston, South Carolina
  - Community Clinical Research, Inc., Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Bayou City Research Limited, Houston, Texas
  - Claghorn-Lesem Research Clinic, Inc, Houston, Texas
  - Mary Ann Knesevich, MD, PA, Irving, Texas
  - InSite Clinical Research, Plano, Texas
  - Frontier Institute, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 500 participants taking antipsychotic drugs: 175 participants in the risperidone cohort, 155 participants in the olanzapine cohort and 170 participants in the aripiprazole cohort were randomized and received study drug in one of two iloperidone treatment arms: gradual switch or immediate switch. 1 randomized participant did not receive study drug.
Period: Overall Study
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Started | 241 (Includes 1 patient randomized in error.) | 260
Safety Population: Received Study Drug | 240 | 260
Completed | 168 | 178
Not Completed | 73 | 82
Not completed — Adverse Event | 25 | 39
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 5 | 4
Not completed — Patient withdrew consent | 14 | 11
Not completed — Lost to Follow-up | 15 | 17
Not completed — Administrative problems | 1 | 1
Not completed — Protocol deviation | 12 | 9
Not completed — Randomized in error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch | Total
Number analyzed (Participants) | 240 | 260 | 500
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline Measures are based on the Safety Population that includes all randomized participants who received study drug.
  years | 42.3 (10.98) | 44.2 (10.92) | 43.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 95 | 165
  Male | 170 | 165 | 335

OUTCOME MEASURES:

1. Primary Outcome: Integrated Clinical Global Impression of Change (I-CGI-C) at Week 12
Description: The I-CGI-C at Week 12 was the overall impression of medically qualified raters using three separate Clinical Global Impression of Change scales: efficacy (E-CGI-C); safety and tolerability (ST-CGI-S); and overall severity (I-CGI-S) combined for a total score. The I-CGI-C scale ranged from 1 to 7 with lower scores indicating improvement (1=very much improved, 2=much improved, 3=minimally improved), higher scores indicating worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicating no change.
Time Frame: Week 12
Population: Participants from the Full Analysis Set (three cohorts combined: risperidone, olanzapine or aripiprazole) with data available for analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 235 | 256
Score on a scale | 2.826 (1.1244) | 2.824 (1.3300)

2. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) at Week 12
Description: The TSQM consisted of 14 questions about the patient's satisfaction with the drug in 4 domains: Effectiveness [3 questions scored as 1(extremely dissatisfied) to 7(extremely satisfied)], Side Effects [question 4 scored as 0(no) or 1(yes);question 5 scored as 1(extremely bothersome) to 5(not at all bothersome);questions 6 - 8 scored as 1(a great deal) to 5(not at all)], Convenience [questions 9 and 10 scored as 1(extremely difficult) to 7 (extremely easy);question 11 scored as 1(extremely inconvenient) to 5 (extremely convenient)] and Global Satisfaction [question 12 scored as 1(not at all confident) to 7(extremely confident);question 13 scored as 1(not at all certain) to 5(extremely certain);question 14 scored as 1(extremely dissatisfied) to 5(extremely satisfied)]. The scores of each of the domains were added together and an algorithm used to create a score of 0 to 100. Higher scores for each domain indicate a better outcome. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Full Analysis Set with data available for analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 214 | 233
Score on a scale
  Change from baseline 3 cohorts combined | 14.1 (29.56) | 12.7 (27.89)
  Change from baseline risperidone cohort (n=75,85) | 14.4 (27.0) | 16.6 (29.65)
  Change from baseline olanzapine cohort (n=70,67) | 13.3 (28.17) | 9.9 (28.60)
  Change from baseline aripiprazole cohort (n=69,81) | 14.8 (33.72) | 11.0 (25.12)

3. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events or Death
Description: Adverse event are defined as any unfavorable and unintended diagnosis, symptoms, sign (including an abnormal lab finding), syndrome or disease which either occurs during the study, having been absent at baseline, or if present at baseline appear to worsen.
  Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization , cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgments of the investigators represent significant hazards.
  Additional information about adverse events can be found in the Adverse Event section.
Time Frame: 12 Weeks
Population: Participants from the Safety Analysis Set- all randomized participants who received study drug (three cohorts combined: risperidone, olanzapine or aripiprazole) with data available for analyses.
Measure: Number; unit: Participants
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 240 | 260
Participants
  Serious Adverse Events | 8 | 7
  Adverse Events | 196 | 207
  Death | 0 | 0

4. Secondary Outcome: Change From Baseline in the Efficacy Clinical Global Impression of Severity (E-CGI-S) at Week 12
Description: Medically qualified raters use the E-CGI-S scale at Baseline and Week 12 to assess the effectiveness of treatment by examining changes in positive symptoms [hallucinations (false perceptions), delusions (false beliefs), paranoia (unfounded distrust), conceptual disorganization (loosening of associations), or hostility], negative symptoms [apathy (lack of interest), avolition (lack of motivation), alogia (poverty of speech), and anhedonia (absence of pleasure)] and cognitive symptoms [concentration difficulties, difficulties with executive function (integrative reasoning), and illogical thinking] in the previous 7 days on a scale of 1 to 7 (1=normal, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill or 7=among the most extremely ill). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Full Analysis Set with data available for analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 235 | 256
Score on a scale
  Change from baseline 3 cohorts combined | -0.8 (0.89) | -0.8 (0.89)
  Change from baseline risperidone cohort (n=81,92) | -0.9 (0.82) | -0.9 (0.85)
  Change from baseline olanzapine cohort (n=77,74) | -0.8 (0.96) | -0.6 (0.88)
  Change from baseline aripiprazole cohort (n=77,90) | -0.8 (0.89) | -0.9 (0.92)

5. Secondary Outcome: Change From Baseline in the Safety and Tolerability Clinical Global Impression of Severity (ST-CGI-S) at Week 12
Description: Medically qualified raters used the ST-CGI-S at Baseline and Week 12 to evaluate safety and tolerability in the previous 7 days on a scale of 1 to 7 (1=Normal-no symptoms, 2=borderline severity, 3=mild impairment, 4=moderate, 5=marked, 6=severe, 7=among the most severe.) A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Full Analysis Set with data available for analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 235 | 256
Score on a scale
  Change from baseline 3 cohorts combined | -0.9 (1.29) | -0.8 (1.45)
  Change from baseline risperidone cohort (n=81,92) | -1.1 (1.27) | -0.9 (1.49)
  Change from baseline olanzapine cohort (n=77,74) | -0.9 (1.20) | -0.9 (1.36)
  Change from baseline aripiprazole cohort (n=77,90) | -0.8 (1.39) | -0.4 (1.45)

6. Secondary Outcome: Change From Baseline in Integrated Clinical Global Impression of Severity (I-CGI-S) at Week 12
Description: I-CGI-S incorporated the overall, combined impression of illness severity based upon the E-CGI-S and ST-CGI-S. Medically qualified raters evaluated the patient's illness in the previous 7 days at Baseline and Week 12 on a scale of 1 to 7 (1=normal not at all ill, 2=borderline mental illness or impairment, 3=mildly ill or impaired, 4=moderately ill or impaired, 5=marked ill or impaired, 6= severely ill or impaired or 7=among the most extremely ill patients. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Number analyzed (Participants) | 235 | 256
Score on a scale
  Change from baseline 3 cohorts combined | -0.9 (0.95) | -0.9 (0.97)
  Change from baseline risperidone cohort (n=81,92) | -0.9 (0.85) | -1.0 (0.89)
  Change from baseline olanzapine cohort (n=77,74) | -0.8 (0.96) | -0.7 (0.98)
  Change from baseline aripiprazole cohort (n=77,80) | -1.0 (1.04) | -0.9 (1.04)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety Set includes all randomized participants who received at least one dose of study drug.
Arm/Group | Iloperidone Gradual Switch | Iloperidone Immediate Switch
Serious Adverse Events (participants affected / at risk) | 8/240 | 7/260
Other Adverse Events (participants affected / at risk) | 148/240 | 155/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone Gradual Switch (N=240) | Iloperidone Immediate Switch (N=260)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Concomitant disease progression (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Social stay hospitalisation (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone Gradual Switch (N=240) | Iloperidone Immediate Switch (N=260)
Dry mouth (Gastrointestinal disorders) | 43 | 54
Nausea (Gastrointestinal disorders) | 13 | 17
Fatigue (General disorders) | 21 | 20
Weight increased (Investigations) | 29 | 20
Increased appetite (Metabolism and nutrition disorders) | 13 | 14
Dizziness (Nervous system disorders) | 42 | 58
Headache (Nervous system disorders) | 17 | 19
Sedation (Nervous system disorders) | 22 | 22
Somnolence (Nervous system disorders) | 34 | 25
Anxiety (Psychiatric disorders) | 11 | 18
Insomnia (Psychiatric disorders) | 20 | 25
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.